CLINICAL TRIAL: NCT06508944
Title: Efficacy of Vaginal 17β-Estradiol on the Urinary Storage Symptoms in Postmenopausal Women: A Randomized Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy of Vaginal 17β-Estradiol on the Urinary Storage Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MURA2024/10; RF_67069 (Other Grant/Funding Number: Faculty of Medicine, Ramathibodi Hospital, MU)
Record Dates: First submitted 2024-07-05; First posted 2024-07-18 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Lower Urinary Tract Symptoms; Female Genitourinary Disease; Urinary Stress Incontinence; Urinary Urge Incontinence; Nocturia; Quality of Life; Voiding Disorders; Vagina Atrophy; Urethral Atrophy; Overactive Bladder; Overactive Bladder Syndrome; Bladder, Overactive
Keywords: 17 beta-estradiol; lower urinary tract symptoms; postmenopause; female genitourinary diseases; urethral maturation index; vaginal pH; ICIQ-FLUTS; ICIQ-LUTSqol; PGI-I; randomized controlled trial; vaginal estrogen; urinary stress incontinence; urinary urge incontinence; nocturia; quality of Life; voiding Disorders; vagina Atrophy; urethral Atrophy; daytime frequency; urgency; behavioral modification; Kegel's exercise; bladder training; bladder diary
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Female Urogenital Diseases; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Nocturia; Urinary Bladder, Overactive | interventions — Estradiol; stearic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Behavioral modifications and vaginal 17beta-estradiol (Experimental): • 17beta-Estradiol 10 mcg + Behavioral modifications
  Interventions: Drug: vaginal 17 beta-estradiol; Behavioral: Behavioral modifications
- Group B: Behavioral modifications + Placebo (Placebo Comparator): • Placebo + Behavioral modifications
  Interventions: Drug: Placebo; Behavioral: Behavioral modifications

INTERVENTIONS:
Drug: vaginal 17 beta-estradiol — * Femiest® Haupt Pharma Munster GMBH, Muenster, Germany
  * The assigned dosage will be one vaginal tablet daily for two weeks then one vaginal tablet twice a week for 10 weeks.
  Other Names: Femiest; ESTRADIOL HEMIHYDRATE; vagifem
  Arms: Group A: Behavioral modifications and vaginal 17beta-estradiol
Drug: Placebo — * Placebo is produced by Chulalongkorn University Drug and Health Products Innovation & Promotion Center.
  * The assigned dosage will be one vaginal tablet daily for two weeks then one vaginal tablet twice a week for 10 weeks.
  Other Names: Agglomerated Lactose; Microcrystalline cellulose PH 102; Magnesium stearate
  Arms: Group B: Behavioral modifications + Placebo
Behavioral: Behavioral modifications — Behavioral modifications for women with storage symptoms of lower urinary tract symptoms (LUTS) involve strategies such as regulating fluid intake, avoiding bladder irritants, practicing bladder training techniques (scheduled and delayed voiding), performing pelvic floor muscle exercises, managing weight, increasing dietary fiber, maintaining a bladder diary, setting a regular voiding schedule, utilizing stress management techniques, and educating patients about LUTS.

SUMMARY:
The goal of this clinical trial is to evaluate whether vaginal 17β-estradiol effectively treats storage symptoms of lower urinary tract symptoms (LUTS) and enhances quality of life. The main questions it aims to answer are:

* What is the efficacy of vaginal 17β-estradiol treatment compared to placebo in alleviating storage symptoms of LUTS?
* How does vaginal 17β-estradiol treatment affect the urethral maturation index and vaginal pH compared to placebo?
* What impact does vaginal 17β-estradiol treatment have on overall quality of life and patients' perception of global improvement (PGI)?

Participants in the trial will undergo the following procedures:

* Screening procedures at the first visit to exclude correctable causes of LUTS and to complete a bladder diary.
* Visit the clinic at 1-2 weeks for a review of the bladder diary and a check-up. Participants will receive the assigned dosage of vaginal 17β-estradiol or placebo: one vaginal tablet daily for two weeks, followed by one vaginal tablet twice a week for 10 weeks.
* The third and fourth visits (at 4 and 12 weeks after treatment) will involve: completion of bladder diaries, questionnaires, vaginal pH testing, collection of urethral maturation index (UMI), observation of intervention's side effects and monitoring of LUTS symptoms.

DETAILED DESCRIPTION:
I. First Visit and Recruitment

Participants will be recruited from the urogynecology clinic, menopause clinic, and urology clinic using hospital and public advertisement. An information sheet in Thai language will be provided to health care providers in the designated outpatient department (OPD) which can ensure the providers convey the correct study information to potential participant. Participants will only be able to enroll into this study one time.

Informed Consent

Individuals with at least one storage symptom of LUTS presenting to clinics in selected OPD will undergo the informed consent process by principal investigator prior to initiating screening procedures. Consent form in Thai language describing in detail the study procedures will be given to the participant privately in a separate room, and extensive discussion of risks and possible benefits of participation in this study will be provided. Participation will be informed that they may withdraw consent at any time throughout the course of this study.

Screening

After documentation of informed consent, principal investigator will interview the participant and perform vital signs and physical examination. The urinalysis will be performed by urinalysis test strip before the start of the study. Screening procedures are as follows;

* Pelvic exam
* Pelvic floor muscle strength measured as Brink scale
* Pelvic Organ Prolapse Quantification (POP-Q), Stress test
* Gynecologic ultrasonography with post-void residual volumes (PVR)
* Urinalysis by urinalysis test strip
* Bladder diary: consecutive three-day diary which the time of each micturition and the volume voided, fluid intake, incontinence episodes, episodes of urgency and sensation will be recorded, as might be the activities performed during or immediately preceding the involuntary loss of urine.

After screening procedure, the appointment will be made for the next visit, which is one or two weeks after first visit.

Bladder diary

The study will incorporate the use of essential diagnostic tool, namely the bladder diary, to assess and monitor the outcomes. These assessments will be administered under the careful supervision of the study investigators. These diagnostic tests play a pivotal role in our research, serving as indispensable instruments for evaluating the progression and ultimate success of the treatment interventions.

II. Second Visit and Randomization

At one or two weeks after 1st visit, the following study procedure will be performed;

* Bladder diary interpretation
* ICIQ-FLUTS questionnaire
* ICIQ-LUTSqol questionnaire
* Vaginal pH
* Urethral maturation index (UMI)

After evaluating all the data collected during the screening process at the initial visit and combining it with the procedures conducted during the second visit, if the woman does not meet all study inclusion or if the woman has an exclusion criterion, she will not be enrolled into this study. A screening log will be kept of all who were evaluated for participation to document who is and is not enrolled and reason for not enrolling in this study.

Women who meet inclusion criteria will be randomized with block randomization technique and a ratio of treatments of 1:1. The sequence generation will be performed under supervision of a senior statistician at the section of Clinical Epidemiology and Biostatistics in Ramathibodi Hospital. The random sequences will be generated using Stata version 18. This is an automated process with no interfere from the investigators. Upon a subject's successful enrollment in the clinical trial following eligibility assessment, principal investigator or research personnel shall provide participants with a comprehensive Thai guidebook for behavior modification which is designed to ensure the harmonization of knowledge and behaviors among all trial participants. This guidebook was developed and published by The International Urogynecological Association (IUGA) and will be distributed by research assistants.

Trial Treatment: Dosage Form, Regimen, Route of Administration

* 17beta-Estradiol 10 mcg (Femiest® Pharma Munster GMBH, Muenster, Germany (ESTRADIOL HEMIHYDRATE 0.0103 milligram, pH 6.94)

  17beta-Estradiol will be administered to group A treatment arm intravaginally. The assigned dosage will be one vaginal tablet daily for two weeks then one vaginal tablet twice a week for 10 weeks. Participants will be carefully monitored for any changes in clinical condition in each follow-up visits using logbook. It is important to clarify that the investigators are not using 17beta-Estradiol (Vagifem®) 25 mcg as the study drug. Although 17beta-Estradiol 25 mcg is frequently mentioned in literature reviews and has been historically used for treating vaginal dryness, this drug is currently not available in Thailand. Therefore, the investigators are using 17beta-Estradiol (Femiest®) 10 mcg as an alternative for our study drug. Notably, 17beta-Estradiol 10 mcg has been shown to provide a therapeutic dose equivalent to that of 17beta-Estradiol 25 mcg for treatment, as stated by the FDA. This decision ensures that participants receive an effective and appropriate dosage while adhering to the availability of medications in our region.
* Placebo

Placebo will be administered to group B treatment arms intravaginally. The assigned dosage will be one vaginal tablet daily for two weeks then one vaginal tablet twice a week for 10 weeks. Participants will be carefully monitored for any changes in clinical condition in each follow-up visits. Placebo is produced by Chulalongkorn University Drug and Health Products Innovation & Promotion Center, Faculty of Pharmaceutical Sciences, Chulalongkorn University. Details for presentation and packing are as follows;

* Appearance: White, round, biconvex with "E" imprint one side
* Weight: 106 - 110 mg
* Hardness: 4.1 - 4.8 kilopond (kp)
* Thickness: 3.26 - 3.3 mm
* Diameter: 6.02 - 6.03 mm
* Disintegration time: 4 min 58sec - 7min 42sec
* pH: 7.18

Placebo contains

1. Agglomerated Lactose
2. Microcrystalline cellulose PH 102
3. Magnesium stearate

Both subject groups will be counseled on potential signs/symptoms of adverse events and post-marketing experience, such as breast pain, peripheral edema, and postmenopausal bleedings. Due to the vaginal administration and minimal systemic absorption, it is unlikely that any clinically relevant drug interactions will occur with 17beta-Estradiol. However, interactions with other locally applied vaginal treatments will be considered and advised to the patients. If a dose is forgotten, participants will be advised that it should be taken as soon as he/she remembers. A double dose should be avoided.

Random allocation

Each participant in the study will receive a prescription for the research drug, an adequate supply to cover a 12-week treatment duration. This drug will be uniformly packaged within identical containers, featuring a unique alphanumeric code and detailed usage instructions on the label, thereby avoiding the inclusion of the original medication name. The data analysis will be performed by a statistician who will be the sole individual privy to the allocation of drug A or drug B to their respective groups. It is essential to note that the statistician will remain unaware of which of the two is the active drug and which is the placebo. Additionally, an independent statistician will maintain a sealed randomization list as a contingency. Allocation will be as follows;

Group A: 17beta-Estradiol 10 mcg (Femiest® Haupt Pharma Munster GMBH, Muenster, Germany (ESTRADIOL HEMIHYDRATE 0.0103 milligram)

Group B: Placebo

III. Third Visit

At four weeks after 2nd visit, the following study procedure will be performed;

* Bladder diary, the participant will be reminded to provide a three-day diary prior to schedule visit date.
* ICIQ-FLUTS questionnaire
* ICIQ-LUTSqol questionnaire
* PGI-I score
* Vaginal pH
* Urethral maturation index (UMI)

Participants will also have clinical evaluation and vital signs measurements evaluated. Compensation for participants will be provided.

IV. Fourth and Final Visit

At eight weeks after 3rd visit, the following study procedure will be performed;

* Pelvic exam
* Pelvic floor muscle strength measured as Brink scale
* Bladder diary, the participant will be reminded to provide a three-day diary prior to schedule visit date.
* ICIQ-FLUTS questionnaire
* ICIQ-LUTSqol questionnaire
* PGI-I score
* Vaginal pH
* Urethral maturation index (UMI)

Participants will also have clinical evaluation and vital signs measurements evaluated. Compensation for participants will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting with storage phase symptom score more than/equal to 1 evaluated by the ICIQ-FLUTS questionnaire in these items

   * Item 2a) nocturia and/or
   * Item 3a) urgency and/or
   * Item 5a) daytime frequency and/or
   * Item 9a) UUI and/or
   * Item 11a) SUI
2. Being natural or surgical menopause for more than 1 year
3. Absence of urinary tract infection or other identifiable cause
4. Not using hormone replacement therapy or any route of estrogen within 4 weeks
5. Never undergone onabotulinumtoxinA therapy, percutaneous tibial nerve stimulation (PTNS), or neuromodulation for overactive bladder (OAB) treatment
6. Willing to adhere to the research protocol and actively participate in the scheduled follow-up appointments as delineated within the framework of this study

Exclusion Criteria:

1. Contraindication for estrogen therapy: undiagnosed abnormal vaginal bleeding, previous thromboembolic event, breast cancer, gynecologic/genitourinary malignancy, active liver disease
2. Pelvic organ prolapse of anterior compartment stage III and IV
3. Immunocompromised patient or taking immunosuppressant drug
4. History of antibiotics drug use within the past 7 days
5. History of bladder outlet obstruction
6. History of using anti-muscarinics, beta3-adrenoceptor agonists, vaginal energy-based devices (laser and radiofrequency) or electromagnetic energy-based therapies within the past 2 weeks
7. History of documented positive urine culture in the past 6 weeks
8. Have an allergic reaction to study's drug
9. Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Storage symptom improvement | The patients were monitored closely for 1 and 3 months after treatment.
  Storage Symptom Improvement: This will be evaluated using the International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), validated in Thai. The questionnaire includes 5 items addressing storage symptoms:
  * 2a) Nocturia
  * 3a) Urgency
  * 5a) Daytime frequency
  * 9a) Urgency urinary incontinence (UUI)
  * 11a) Stress urinary incontinence (SUI)
  Each severity item is rated from 0 to 4, and each bothersome item from 0 to 10. The total severity score ranges from 0 to 20, and the total bothersome score ranges from 0 to 50. Higher scores indicate worse outcomes.
  Outcome Interpretation:
  * Improved: Mean ICIQ-FLUTS post-treatment score < pre-treatment score.
  * Not Improved: Mean ICIQ-FLUTS post-treatment score ≥ pre-treatment score.

SECONDARY OUTCOMES:
The impact of urinary storage symptoms on quality of life | The patients were monitored closely for 1 and 3 months after treatment.
  • Assess the impact of urinary storage symptoms on quality of life with reference to social effects by Thai version of International Consultation on Incontinence Questionnaire Urinary Incontinence Quality of Life (ICIQ-LUTSqol), which comprises 20 items. The ranges from 19 to 76, with greater values indicating increased impact on quality of life. ICIQ-LUTSqol is a validated Thai adaptation of King's Health Questionnaire (KHQ).
Global Improvement score | The patients were monitored closely for 1 and 3 months after treatment.
  The Global Improvement score is evaluated using the Thai version of the Patient Global Impression of Improvement (PGI-I) scale. This scale is a widely used, patient-reported measure that assesses the patient's overall perception of improvement following a treatment. The PGI-I is typically rated on a 7-point scale, where the minimum value is 1 and the maximum value is 7. On this scale, a score of 1 indicates that the patient feels "very much improved," while a score of 7 indicates that the patient feels "very much worse." Therefore, lower scores on the PGI-I represent better outcomes, reflecting greater improvement in the patient's condition, while higher scores denote worse outcomes, indicating little to no improvement or a decline in the patient's condition.
Urethral maturation index (UMI) and maturation value (MV) | The patients were monitored closely for 1 and 3 months after treatment.
  We will use wet cotton buds coated with normal saline solution (NSS) to gently swab the distal urethra for cytologic preparation. Smear slides will be prepared for cytologic evaluation by immediately immersing them in 95% alcohol for 24 hours and staining them with a Papanicolaou stain. The urethral epithelial cell will be examined under a microscope and classified into three types: parabasal cells, intermediate cells, and superficial cells by an independent cytologist. Two hundred cells were counted at each high-power field which was randomly chosen. Six high-power fields were evaluated and the mean of the cell numbers was calculated. MV is a derived value from the proportion of different cell types and is, therefore, unitless.
  Maturation value (MV) = (% parabasal cells × 0) + (% intermediate cells × 0.5) + (% superficial cells × 1.0)
  Interpretation:
  * MV = 0-49 will indicate low estrogen effect
  * MV = 50-64 = moderate estrogen effect
  * MV = 65-100 = high estrogen effect
Vaginal pH | The patients were monitored closely for 1 and 3 months after treatment.
  To assess pH, a piece of litmus paper (MQuant® pH-indicator stripe) will be placed on the lateral vaginal wall until moistened. A pH of 4.6 or greater indicates vulvovaginal atrophy (VVA)(31). According to a preliminary double-blinded study in 67 symptomatic postmenopausal women confirmed that atrophic vaginitis is associated with an increase in the lateral wall vaginal pH and this finding is paralleled by similar changes in pH in the urethra. Also, locally applied vaginal conjugated estrogen cream can normalizes the pH in the vagina and urethra Thus, the testing of the vaginal pH serves both as a surrogate for evaluating urethral pH and as a monitor of compliance with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pornthip Harncharoenkul, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomaszewski J. Postmenopausal overactive bladder. Prz Menopauzalny. 2014 Dec;13(6):313-29. doi: 10.5114/pm.2014.47984. Epub 2014 Dec 30. PMID 26327873
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Weber MA, Kleijn MH, Langendam M, Limpens J, Heineman MJ, Roovers JP. Local Oestrogen for Pelvic Floor Disorders: A Systematic Review. PLoS One. 2015 Sep 18;10(9):e0136265. doi: 10.1371/journal.pone.0136265. eCollection 2015. PMID 26383760
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Iosif CS, Batra S, Ek A, Astedt B. Estrogen receptors in the human female lower uninary tract. Am J Obstet Gynecol. 1981 Dec 1;141(7):817-20. doi: 10.1016/0002-9378(81)90710-9. PMID 7198384
- [Background] Chung da J, Bai SW. Roles of sex steroid receptors and cell cycle regulation in pathogenesis of pelvic organ prolapse. Curr Opin Obstet Gynecol. 2006 Oct;18(5):551-4. doi: 10.1097/01.gco.0000242959.63362.1e. PMID 16932051
- [Background] Rud T, Andersson KE, Asmussen M, Hunting A, Ulmsten U. Factors maintaining the intraurethral pressure in women. Invest Urol. 1980 Jan;17(4):343-7. PMID 7188694
- [Background] Matsubara S, Okada H, Shirakawa T, Gotoh A, Kuno T, Kamidono S. Estrogen levels influence beta-3-adrenoceptor-mediated relaxation of the female rat detrusor muscle. Urology. 2002 Apr;59(4):621-5. doi: 10.1016/s0090-4295(01)01583-7. PMID 11927339
- [Background] Shenfeld OZ, McCammon KA, Blackmore PF, Ratz PH. Rapid effects of estrogen and progesterone on tone and spontaneous rhythmic contractions of the rabbit bladder. Urol Res. 1999 Oct;27(5):386-92. doi: 10.1007/s002400050168. PMID 10550529
- [Background] Peyronnet B, Mironska E, Chapple C, Cardozo L, Oelke M, Dmochowski R, Amarenco G, Game X, Kirby R, Van Der Aa F, Cornu JN. A Comprehensive Review of Overactive Bladder Pathophysiology: On the Way to Tailored Treatment. Eur Urol. 2019 Jun;75(6):988-1000. doi: 10.1016/j.eururo.2019.02.038. Epub 2019 Mar 26. PMID 30922690
- [Background] Chen HY, Lin YN, Chen WC, Wang SJ, Chen CJ, Chen YH. Urethral proteomic analysis in ovariectomized mice administered 17beta-oestradiol replacement therapy. J Obstet Gynaecol. 2017 Aug;37(6):757-765. doi: 10.1080/01443615.2017.1292225. Epub 2017 Mar 28. PMID 28350532
- [Background] Johnston SL. Pelvic floor dysfunction in midlife women. Climacteric. 2019 Jun;22(3):270-276. doi: 10.1080/13697137.2019.1568402. Epub 2019 Mar 11. PMID 30857432
- [Background] Benness C, Wise BG, Cutner A, et al. Does low dose vaginal oestradiol improve frequency and urgency in postmenopausal women. Int Urogynaecol J. 1992;3:281.
- [Background] Eriksen PS, Rasmussen H. Low-dose 17 beta-estradiol vaginal tablets in the treatment of atrophic vaginitis: a double-blind placebo controlled study. Eur J Obstet Gynecol Reprod Biol. 1992 Apr 21;44(2):137-44. doi: 10.1016/0028-2243(92)90059-8. PMID 1587379
- [Background] Pratt TS, Suskind AM. Management of Overactive Bladder in Older Women. Curr Urol Rep. 2018 Sep 10;19(11):92. doi: 10.1007/s11934-018-0845-5. PMID 30203368
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Titapant V, Ek-anankul W, Chawanpaiboon S. Prevalence of Overactive Bladder Among Nurses at Siriraj Hospital. Siriraj Med J. 2002 Nov. 1;54(11):710-5.
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Robinson D, Cardozo L. Estrogens and the lower urinary tract. Neurourol Urodyn. 2011 Jun;30(5):754-7. doi: 10.1002/nau.21106. PMID 21661025
- [Background] Artibani W. Complications of surgery for stress incontinence. In: Cardozo L, Staskin L, editors. Textbook of female urology and urogynecology. 2nd ed. Taylor & Francis Ltd; 2007;1345-62.
- [Background] Cardozo L., Staskin, D. (Eds.). Textbook of Female Urology and Urogynecology: Clinical Perspectives (5th ed.). Boca Raton: CRC Press; 2023
- [Background] Simunic V, Banovic I, Ciglar S, Jeren L, Pavicic Baldani D, Sprem M. Local estrogen treatment in patients with urogenital symptoms. Int J Gynaecol Obstet. 2003 Aug;82(2):187-97. doi: 10.1016/s0020-7292(03)00200-5. PMID 12873780
- [Background] Cardozo LD, Wise BG, Benness CJ. Vaginal oestradiol for the treatment of lower urinary tract symptoms in postmenopausal women--a double-blind placebo-controlled study. J Obstet Gynaecol. 2001 Jul;21(4):383-5. doi: 10.1080/01443610120059941. PMID 12521832
- [Background] Mostafaei H, Janisch F, Mori K, Quhal F, Pradere B, Hajebrahimi S, Roehrborn CG, Shariat SF. Placebo Response in Patients with Oral Therapy for Overactive Bladder: A Systematic Review and Meta-analysis. Eur Urol Focus. 2022 Jan;8(1):239-252. doi: 10.1016/j.euf.2021.02.005. Epub 2021 Mar 3. PMID 33674256
- [Background] Cardozo L, Rovner E, Wagg A, Wein A, Abrams P. (Eds) Incontinence 7th Edition. Bristol UK: ICI-ICS. International Continence Society. 2023.
- [Background] Mostafaei H, Mori K, Quhal F, Miura N, Motlagh RS, Pradere B, Laukhtina E, Lysenko I, Ghaffari S, Hajebrahimi S, Shariat SF. Nocebo Response in the Pharmacological Management of Overactive Bladder: A Systematic Review and Meta-analysis. Eur Urol Focus. 2021 Sep;7(5):1143-1156. doi: 10.1016/j.euf.2020.10.010. Epub 2020 Nov 3. PMID 33153953
- [Background] Chattrakulchai K, Manonai J, Silpakit C, Wattanayingcharoenchai R. Validation of the Thai version of the International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS). Int Urogynecol J. 2020 Dec;31(12):2603-2610. doi: 10.1007/s00192-020-04422-1. Epub 2020 Jul 4. PMID 32620979
- [Background] Kochakarn W, Pummangura N, Kijvikai K, Viseshsindh W, Sukying C, Lertsithichai P. Reliability of a Thai version of King's Health Questionnaire in Thai females with overactive bladder symptoms. J Med Assoc Thai. 2005 Nov;88(11):1526-34. PMID 16471097
- [Background] Srikrishna S, Robinson D, Cardozo L. Validation of the Patient Global Impression of Improvement (PGI-I) for urogenital prolapse. Int Urogynecol J. 2010 May;21(5):523-8. doi: 10.1007/s00192-009-1069-5. Epub 2009 Dec 15. PMID 20013110
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Mension E, Alonso I, Tortajada M, Matas I, Gomez S, Ribera L, Ros C, Angles-Acedo S, Castelo-Branco C. Genitourinary Syndrome of Menopause Assessment Tools. J Midlife Health. 2021 Apr-Jun;12(2):99-102. doi: 10.4103/jmh.jmh_93_21. Epub 2021 Jul 27. PMID 34526742
- [Background] Notelovitz M. Estrogen therapy in the management of problems associated with urogenital ageing: a simple diagnostic test and the effect of the route of hormone administration. Maturitas. 1995 Dec;22 Suppl:S31-3. doi: 10.1016/0378-5122(95)00960-4. PMID 8775774
- [Background] Manonai J. Management of Female Urogenital Atrophy. 1st ed. Bangkok: Ramathibodi Press; 2014:52-3.
- [Background] Manonai J, Seif C, Bohler G, Junemann KP. The effect of Pueraria mirifica on cytologic and urodynamic findings in ovariectomized rats. Menopause. 2009 Mar-Apr;16(2):350-6. doi: 10.1097/gme.0b013e318188b279. PMID 19098688
- [Background] Bergman A, Karram MM, Bhatia NN. Changes in urethral cytology following estrogen administration. Gynecol Obstet Invest. 1990;29(3):211-3. doi: 10.1159/000293384. PMID 2358196
- [Background] Simon JA, Reape KZ, Wininger S, Hait H. Randomized, multicenter, double-blind, placebo-controlled trial to evaluate the efficacy and safety of synthetic conjugated estrogens B for the treatment of vulvovaginal atrophy in healthy postmenopausal women. Fertil Steril. 2008 Oct;90(4):1132-8. doi: 10.1016/j.fertnstert.2007.07.1359. Epub 2007 Dec 3. PMID 18053998
- [Background] Meisels A. The maturation value. Acta Cytol. 1967 Jul-Aug;11(4):249. No abstract available. PMID 5233434
- [Background] Brunzel NA. Fundamentals of Urine and Body Fluid Analysis. 4 th ed. St.Loius: Elsevier; 2018.
- [Background] Simon J, Nachtigall L, Gut R, Lang E, Archer DF, Utian W. Effective treatment of vaginal atrophy with an ultra-low-dose estradiol vaginal tablet. Obstet Gynecol. 2008 Nov;112(5):1053-60. doi: 10.1097/AOG.0b013e31818aa7c3. PMID 18978105

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT06508944/Prot_SAP_000.pdf